CLINICAL TRIAL: NCT02962700
Title: Effects of Continuous Haemofiltration vs Intermittent Haemodialysis on Microcirculatory Parameters in Septic Shock
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Military Hospital of Tunis (Other)
Responsible Party: Principal Investigator, Hajjej Zied, Doctor, Military Hospital of Tunis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: CVVHFmicro
Record Dates: First submitted 2016-11-04; First posted 2016-11-11 (Estimated); Last update posted 2016-11-11 (Estimated); Status verified 2016-11

CONDITIONS: Septic Shock
Keywords: continuous haemofiltration; intermittent haemodialysis
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CVVHF (Experimental): CVVHF for 48 h interstitial tissue concentrations of lactate, pyruvate, glucose and glycerol were obtained at baseline, 6, 12,18 and 24 hours after initiation of renal replacement by using muscle microdialysis.
  Interventions: Device: muscle microdialysis
- IHD for 4 hours (Active Comparator): Intermittent haemodialysis was carried out during the first 4 h at day 1 and day 2 of the study period.
  Interstitial tissue concentrations of lactate, pyruvate, glucose and glycerol were obtained at baseline, 6, 12,18 and 24 hours after initiation of renal replacement by using muscle microdialysis.
  Interventions: Device: muscle microdialysis

INTERVENTIONS:
Device: muscle microdialysis — Systemic haemodynamics and interstitial tissue concentrations of lactate, pyruvate, glucose and glycerol were obtained at baseline, 6, 12,18 and 24 hours after initiation of renal replacement by using muscle microdialysis.

SUMMARY:
The aim of the study was to investigate whether CVVH, in comparison to intermittent haemodialysis (IHD), is able to improve regional perfusion in septic shock patients studied by muscle microdialysis

DETAILED DESCRIPTION:
A prospective, randomized, clinical study ,including septic shock patients with acute renal failure, aged over 16 years. Patients were randomized to receive either CVVH or IHD for renal replacement therapy. Intermittent haemodialysis was carried out during the first 4 h at day 1 and day 2 of the study period. Systemic haemodynamics and interstitial tissue concentrations of lactate, pyruvate, glucose and glycerol were obtained at baseline, 6, 12,18 and 24 hours after initiation of renal replacement by using muscle microdialysis.

ELIGIBILITY:
Inclusion Criteria:

* septic shock

Exclusion Criteria:

-

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
changes in the concentration of glucose (mmol/l) in the extracellular fluid of the skeletal muscle using a microdialysis probe inserted into the quadriceps femoris muscle. | at baseline, 6, 12, 18, 24, 30, 36, 42 and 48 hours after initiation of renal replacement
changes in the concentration of lactate (mmol/l) in the extracellular fluid of the skeletal muscle using a microdialysis probe inserted into the quadriceps femoris muscle | at baseline, 6, 12, 18, 24, 30, 36, 42 and 48 hours after initiation of renal replacement
changes in the concentration of pyruvate (µmol/l) in the extracellular fluid of the skeletal muscle using a microdialysis probe inserted into the quadriceps femoris muscle | at baseline, 6, 12, 18, 24, 30, 36, 42 and 48 hours after initiation of renal replacement
changes in the concentration of glycerol (µmol/l) in the extracellular fluid of the skeletal muscle using a microdialysis probe inserted into the quadriceps femoris muscle | at baseline, 6, 12,18, 24, 30, 36, 42 and 48 hours after initiation of renal replacement

SECONDARY OUTCOMES:
changes in mean arterial blood pressure | at baseline, 6, 12, 18, 24, 30, 36, 42 and 48 hours after initiation of renal replacement
changes in heart rate | at baseline, 6, 12, 18, 24, 30, 36, 42 and 48 hours after initiation of renal replacement
changes in vasopressor support doses | at baseline, 6, 12, 18, 24, 30, 36, 42 and 48 hours after initiation of renal replacement

CONTACTS AND LOCATIONS:
Overall Officials: mustapha ferhjani, Study Director — Department of C ritical C are Medicine and Anesthesiology, Military Hospital of Tunis, Tunisia, Tunis, Tunisia
Locations (1):
- Military Hopital of Tunis, Tunis, Tunisia